CLINICAL TRIAL: NCT04082936
Title: A Phase 1/2 Open-label, Multicenter Study Evaluating the Safety and Pharmacokinetics of Imvotamab (IGM-2323) as a Single Agent and in Combination in Subjects With Relapsed/Refractory Non-Hodgkin Lymphomas
Brief Title: A Study of Imvotamab Monotherapy and in Combination in Subjects With Relapsed/Refractory Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic Pipeline Prioritization: Clinical development of imvotamab in autoimmune diseases prioritized.
Sponsor: IGM Biosciences, Inc. (Industry)
Collaborators: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IGM-2323-001
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Non-Hodgkin Lymphoma; Follicular Lymphoma; DLBCL; Mantle Cell Lymphoma; Marginal Zone Lymphoma
Keywords: Lymphoma; Non-Hodgkin Lymphoma; DLBCL; Follicular Lymphoma; relapsed or refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1a (Dose Escalation) (Experimental): Subjects will receive imvotamab via intravenous (IV) infusion weekly. No longer enrolling.
  Interventions: Drug: imvotamab
- Phase 1a (Q3W) (Experimental): Subjects will receive imvotamab via intravenous (IV) infusion every 3 weeks. No longer enrolling.
  Interventions: Drug: imvotamab
- Phase 1a (Prior bi-specific) (Experimental): Subjects treated with prior bi-specifics will receive imvotamab via IV infusion weekly. No longer enrolling.
  Interventions: Drug: imvotamab
- Phase 2 (DLBCL) (Experimental): DLBCL subjects will receive imvotamab via IV infusion at a dose and schedule to be determined after reviewing all available response and safety data. No longer enrolling.
  Interventions: Drug: imvotamab
- Phase 2 (FL) (Experimental): FL subjects will receive imvotamab via IV infusion at a dose and schedule to be determined after reviewing all available response and safety data. No longer enrolling.
  Interventions: Drug: imvotamab
- Phase 1b (Combination) (Experimental): Subjects will receive imvotamab via IV infusion weekly and loncastuximab tesirine via IV infusion every 3 weeks.
  Interventions: Drug: imvotamab

INTERVENTIONS:
Drug: imvotamab — Subjects with r/r B-cell NHL will receive IGM-2323 via IV infusion.

SUMMARY:
This is a Phase 1/2 study of imvotamab in adult subjects with relapsed or refractory B-cell Non-Hodgkin Lymphoma. This study will consist of a dose-escalation stage, a combination stage, and a randomized dose-expansion stage where subjects will be enrolled into indication-specific expansion cohorts. imvotamab will be administered intravenously (IV).

Additional CD20-positive NHL histologies (e.g. MZL and MCL), may be allowed with Medical Monitor approval during the Dose-Escalation Phase of the study.

DETAILED DESCRIPTION:
Imvotamab is an engineered bispecific IgM antibody for the treatment of patients with CD20-positive cancers. It contains ten high affinity binding domains for CD20, and one binding domain for CD3. Imvotamab is able to eliminate CD20-positive lymphoma cells by engaging T-cells and lymphoma cells, leading to T-cell dependent cellular cytotoxicity. Additionally, imvotamab is also able to eliminate lymphoma cells by recruiting complement to the surface of lymphoma cells, leading to complement dependent cytotoxicity.

In our preclinical studies, we observed activity against rituximab resistant cells carrying low levels of CD20. We have also observed much lower cytokine release with imvotamab relative to comparable IgG format bispecific T-cell engaging antibodies, which is expected to result in reduced risk of the serious adverse effects from cytokine release syndrome (CRS).

For the combination stage, imvotamab will be combined with loncastuximab tesirine, a CD19-targeting antibody drug conjugate.

ELIGIBILITY:
Key Inclusion Criteria:

* > 18 years of age: ECOG PS 0 or 1
* Relapsed or Refractory Follicular Lymphoma (FL), and Diffuse Large B-cell Lymphoma (DLBCL), Mantle cell Lymphoma (MCL), Marginal Zone Lymphoma (MZL) in dose escalation
* Relapsed or refractory to at least two prior systemic treatment regimens (must include anti-CD20 chemo-immunotherapy regimen). FL/MZL may be enrolled with a least 2 prior systemic regimens which must include an anti-CD20, without the need for a prior chemotherapy regimen)
* At least one bi-dimensionally measurable lesion (>1.5cm in it's longest dimension by computerized tomography (CT scan)
* Good organ function
* Not eligible for autologous stem cell transplant (DLBCL subjects), due to chemoresistant disease, medically unfit (organ function), or unwilling.

Key Exclusion Criteria:

* Prior allogeneic transplant
* ASCT within 100 days prior to the first imvotamab administration.
* Lack of response to prior treatment with CAR-T therapy, subjects with less than 3 months from prior CAR-T therapy to first dose of imvotamab, and prior CAR-T therapy only allowed with Medical Monitor approval.
* Concurrent serious co-morbidities that could limit patients full participation and compliance.
* Prior CD-targeting bispecific antibodies.
* Prior loncastuximab tesirine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Overall Frequency of Adverse Events | Baseline through approximately 30 days after last study treatment
  Percentage of Adverse Events
Overall Response Rate (ORR) | Baseline up to 5 years
  Percentage of measurable disease in subjects who have achieved either complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline up to 5 years
  Percentage of measurable disease in subjects who have achieved either complete response (CR) or partial response (PR)
Duration of Response (DOR) | Baseline up to 5 years
  measured from time of initial response until documented tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: IGM Biosciences, Study Director — IGM Biosciences, Inc.
Locations (26):
- United States (9):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - NYU, New York, New York
  - MSKCC, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutch, Seattle, Washington
- Australia (3):
  - Monash Health, Clayton, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Linear Clinical Resaerch, Nedlands, Western Australia
- Fakultní nemocnice Královské Vinohrady, Prague, Czechia
- France (2):
  - CHU de Poitiers, Poitiers
  - Gustave Roussy, Villejuif
- Italy (3):
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma, RM
  - Azienda Ospedaliero Universitaria di Bologna-Ematologia Bologna, Bologna
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - START-Madrid: Fundacion Jimenez Diaz, Madrid
  - START-Madrid: Centro Integral Oncologico Clara Campal, Madrid